CLINICAL TRIAL: NCT06855914
Title: Outcomes of Surgical Management of Aneurysmal Arteriovenous Fistula in Hemodialysis Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, abanoub saad anis, Principal investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: surgery in aneurysmal AVF
Record Dates: First submitted 2025-02-02; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Arteriovenous Fistula Patency

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- surgical repair (Experimental): surgical repair of AVF
  Interventions: Procedure: surgerical repair

INTERVENTIONS:
Procedure: surgerical repair — surgical repair of AVF aneurysm

SUMMARY:
To evaluate the success rate and patency after surgical management of Arteriovenous fistulas aneurysms

DETAILED DESCRIPTION:
End-stage renal failure is a disease that can affect all organs. The increasing prevalence of afﬂuent-society diseases such as obesity, diabetes, hypertension, or atherosclerosis means that the number of patients diagnosed with end-stage renal disease is systematically growing . Worldwide, the number of patients receiving hemodialysis is estimated at more than 1.4 million, with the annual incident rate growing to 8%, prevalence of ESRD in Egypt raised to 483 patients per million. A well-functioning vascular access is a mainstay to perform an efficient haemodialysis . AVF, described by Brescia and Cimino, remains the first choice for chronic Haemodialysis . It is the best access for longevity and has the lowest association with morbidity and mortality, and for this reason AVF use is strongly recommended by guidelines from different countries . The most common complications of fistulae for HD are lymphedema, infection, aneurysm, stenosis, congestive heart failure, steal syndrome, ischemic neuropathy and thrombosis. It is important to gain information about early clinical symptoms of AVF dysfunction in order to prevent and adequately treat potential complications . Arteriovenous fistula aneurysms are defined by an expansion of the intimal, medial and adventitial layers of the vessel wall to a diameter of more than 18 mm. Aneurysmal degeneration of the venous component of surgically created arteriovenous fistulae (AVFs) is a common clinical finding. prevalence rates ranging widely between 6% and 51% depending on criteria. Although arteriovenous fistula aneurysms (AVFAs) can be prone to thrombosis and can cause cosmetic dissatisfaction, the most catastrophic complication is life-threatening haemorrhage . The decision for surgical intervention relies on the risk of perforation, ulceration, bleeding, and size of aneurysm which leaves a limited space for puncture. The surgical modalities include excision of the aneurysm and primary repair, excision of the aneurysm and interposition graft , repair by end-to-end anastomosis, ligation .

ELIGIBILITY:
Inclusion Criteria:

* All patients with pseudo-aneurysms over AVF
* skin Changes ( Ulceration - Inflammation -Necrosis)
* Huge Enlargement with lack of potential site of Cannulation
* Impending thrombosis of the fistula
* Risk of infection and impending rupture
* Significant Cosmetic concerns causing distress to the patient

Exclusion Criteria:

* Bad general condition, patient with severe comorbidities
* Thrombosed AV fistula
* Age < 18 years
* Anastomotic aneurysms
* Venous Hypertension over AVF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-02-25 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
evaluate patency after surgical repair | baseline
  evaluate patency after surgical repair of aneurysmal arteriovenous fistula
evaluate success rate after repair | baseline
  success rate of surgical repair of aneurysm and can use fistula for further dialysis or not

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Stolic R. Most important chronic complications of arteriovenous fistulas for hemodialysis. Med Princ Pract. 2013;22(3):220-8. doi: 10.1159/000343669. Epub 2012 Nov 2. PMID 23128647
- [Background] Santoro D, Benedetto F, Mondello P, Pipito N, Barilla D, Spinelli F, Ricciardi CA, Cernaro V, Buemi M. Vascular access for hemodialysis: current perspectives. Int J Nephrol Renovasc Dis. 2014 Jul 8;7:281-94. doi: 10.2147/IJNRD.S46643. eCollection 2014. PMID 25045278
- [Background] 2. Abdel-Fattah El-Ballat M, Ahmed El-Sayed M, Kamel Abdel-Raouf Emam H. Epidemiology of End Stage Renal Disease Patients on Regular Hemodialysis in El-Beheira Governorate, Egypt. Vol. 76, The Egyptian Journal of Hospital Medicine. 2019.
- [Background] Plonski A, Plonski AF, Glowinski J. Surgical Management, Prevention and Outcomes for Aneurysms of Arteriovenous Dialysis Fistulas: A Case Series Study and Review. Int J Environ Res Public Health. 2023 Jun 29;20(13):6256. doi: 10.3390/ijerph20136256. PMID 37444103